CLINICAL TRIAL: NCT03259126
Title: Evaluation of a New Device Placed Under the Angiographic Table to Reduce Operator Radiation Exposure During Percutaneous Coronary Procedures Through Transradial Approach
Brief Title: EXTended pRotective Curtain Under Table to Reduce Operator RAdiation Dose in Percutaneous Coronary Procedures
Acronym: EXTRA-RAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Sandro Pertini, Roma (Other)
Responsible Party: Principal Investigator, Alessandro Sciahbasi, MD, MD, PhD, Ospedale Sandro Pertini, Roma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pertini05
Record Dates: First submitted 2017-08-16; First posted 2017-08-23 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Radiation; X-rays; Effects; Coronary Disease
Keywords: Transradial; Coronary; X-ray; Radiation; Curtain
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: Comparison of operator radiation dose at pelvic level during percutaneous coronary procedures through transradial access with or without an extension of the leaded curtain under table
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCUT (Experimental): Use of a "Small Curtain under table" (SCUT) placed under the cranial part of the angiographic table
  Interventions: Device: SCUT
- Control (No Intervention): Control Group without the SCUT

INTERVENTIONS:
Device: SCUT — Two different home made curtains were attached to the angiographic table
  Arms: SCUT

SUMMARY:
Radiation dose to interventional cardiologists performing transradial percutaneous coronary procedures is higher compared to those performing transfemoral exams. The radiation dose seems particularly high at pelvic level. We prepared an home-made protective extension of the leaded curtain under table that should reduce the operator exposure during interventional coronary procedures. The aim of the study is to evaluate the procedural efficacy of the protective extension on the operator radiation dose at pelvic level

DETAILED DESCRIPTION:
Interventional cardiologists are routinely exposed to x-rays during their activity increasing the risk of deterministic and stochastic effects. Consequently all the operators should be aware of the possible risks and they should apply all efforts to reduce the radiation dose according to the "As Low As Reasonably Achievable" (ALARA) principle. Moreover interventional cardiologists have to utilise adequate protection devices (lead apron, protective thyroid collar, lead glasses).

Operator performing transradial access procedures showed a significantly higher radiation exposure compared to those performing transfemoral interventions. So, transradial operators should use adjunctive protective shields (as leaded pelvic drapes placed on the patient abdomen) in order to reduce their radio-exposition.

During transradial access a particularly high radiation exposure is observed at operator pelvic level and the use of the protective adjunctive drapes placed on the patient abdomen is only partially effective to control this exposition.

Aim of our study was to evaluate the effect of a protective extension of the leaded curtain placed under the angiographic table in term of operator radiation exposure at pelvic level

ELIGIBILITY:
Inclusion Criteria:

all patient undergoing percutaneous coronary procedures through transradial access

Exclusion Criteria:

1. Interventions performed through a different vascular access
2. Procedures performed in patients with ST elevation acute myocardial infarction
3. Haemodynamic instability
4. Lack of written informed consent
5. Age < 18 years old
6. Previous coronary artery by-pass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Operator pelvic dose | 24 hours
  Operator radiation dose at pelvic level

SECONDARY OUTCOMES:
Operator thorax dose | 24 hours
  Operator radiation dose at thorax level
Operator head dose | 24 hours
  Operator radiation dose at head level
Operator pelvic dose and experimental curtain utilized | 24 hours
  Operator radiation Dose at pelvic level comparing the two different experimental leaded curtain utilized

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sciahbasi, MD, PhD, Principal Investigator — Ospeadale Sandro Pertini ASL RM2
Locations (1):
- Ospedale Sandro Pertini, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sciahbasi A, Sarandrea A, Rigattieri S, Patrizi R, Cera M, Di Russo C, Zezza L, Fedele S, Ferraiuolo G. Extended Protective Shield Under Table to Reduce Operator Radiation Dose in Percutaneous Coronary Procedures. Circ Cardiovasc Interv. 2019 Feb;12(2):e007586. doi: 10.1161/CIRCINTERVENTIONS.118.007586. PMID 30732471